CLINICAL TRIAL: NCT01951352
Title: Effects of Surfactants on the Innate Immune System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tissa Hata, MD, MD, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UCSD 111295
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: study; meant; individuals
MeSH Terms: interventions — Soaps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Soap recipient (Experimental): The forearms of all subjects will eventually be washed with the same soaps. There is only one arm for this study.
  Interventions: Other: Soap

INTERVENTIONS:
Other: Soap

SUMMARY:
In this study we will test the ability of different commercially available hand soaps to effect the amount of anti-microbial peptides present on the surface of the human skin after washing with these soaps. Based on our experiments on pig skin, we expect the amount of antimicrobial peptide expression to decrease after using these different soaps.

DETAILED DESCRIPTION:
We will use tape-stripping methods to determine the level of antimicrobial peptides (specifically LL-37) present on the human skin after washing with different commercially available hand soaps. First we will do a baseline tape-stripping procedure to measure the amount of LL-37 on subjects' forearms. Tape stripping involves applying small, round tapes (CuDerm, Dallas, TX) to the skin, massaging them for about 10 second, and then removing them. This process is repeated 9 times for each tape. After doing baseline tape stripping samples, each participant's forearms will be washed with a different soap. The soap will be rinsed off, and the skin allowed to dry. After the forearms are dry (about 5 minutes later), repeat tape-stripping will be performed. This tape-stripping process will then be repeated 4 hours later, and then 24 hours later as well. Results of the LL-37 expression at each time point will then be compared between soaps.

ELIGIBILITY:
Inclusion Criteria:

Those who meet all of the following criteria are eligible for enrollment into the study:

1. Age 18-60 years
2. Male or female of any race and ethnicity
3. Subject agrees to comply with study requirements.

Exclusion Criteria:

1. Subjects with severe medical condition(s) that in the view of the investigator prohibits participation in the study
2. Dermatologic disease such as psoriasis or atopic dermatitis which may have inherently abnormal antimicrobial peptide levels
3. Subject has Netherton's syndrome or other genodermatoses that result in a defective epidermal barrier
4. Pregnant or nursing females
5. Immunocompromised subjects (e.g., lymphoma, HIV/AIDS, Wiskott-Aldrich Syndrome), or with a history of active or malignant disease (excluding non-melanoma skin cancer) as determined by the participant's medical history.
6. Subjects with a history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol
7. Subjects with significant concurrent medical condition(s) at screening that in the view of the investigator prohibits participation in the study (e.g., severe concurrent allergic disease, condition associated with malignancy, and condition associated with immunosuppression)
8. Active viral or fungal skin infections at the target areas
9. Previous participation in this study
10. Ongoing participation in an investigational drug trial
11. Use of any oral or topical antibiotic during the study and up to one week prior to entering the study
12. Use of any local topical medications less than one week prior to screening
13. Use of any systemic immunosuppressive therapy less than four weeks prior to screening.
14. Subjects with a history of or propensity to developing reactions after use of over the counter cleansers
15. History of allergy to adhesive tape

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Division of Dermatology, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Soap Recipient: The forearms of all subjects will eventually be washed with the same soaps. There is only one arm for this study.
  Soap
Period: Overall Study
Arm/Group | Soap Recipient
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Soap Recipient
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Normalized LL-37 Expression
Description: LL-37 expression was measured using tape-stripping methods and expressed relative to baseline.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Soap Recipient
Number analyzed (Participants) | 10
percentage of baseline | 100 (0)

2. Primary Outcome: Normalized LL-37 Expression
Description: LL-37 was measured using tape-stripping methods and is expressed relative to baseline levels
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Soap Recipient
Number analyzed (Participants) | 10
percentage of baseline | 82 (10)

3. Primary Outcome: Normalized LL-37 Expression
Description: LL-37 expression was measured using tape-stripping methods and expressed relative to baseline.
Time Frame: 5 minutes
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Soap Recipient
Number analyzed (Participants) | 10
percentage of baseline | 77 (30)

4. Primary Outcome: Normalized LL-37 Expression
Description: LL-37 expression was measured using tape-stripping methods and expressed relative to baseline.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: percentage of baseline
Arm/Group | Soap Recipient
Number analyzed (Participants) | 10
percentage of baseline | 87 (20)

ADVERSE EVENTS:
Arm/Group | Soap Recipient
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No